CLINICAL TRIAL: NCT04407533
Title: Dietary Intake and Eating Habits During the COVID-19 Pandemic
Acronym: COVIDiet
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Stéphanie Chevalier, Associate Professor, McGill University
Other Study IDs: 20-04-064
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: COVID-19
Keywords: nutrition; dietary intake; eating habits; lifestyle behaviours; physical activity; sleep; artificial intelligence; mobile application
MeSH Terms: conditions — COVID-19; Feeding Behavior; Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Diet tracking and survey — Mobile AI-based food diary application and online questionnaires

SUMMARY:
The COVID-19 pandemic affects eating habits, diet quality and physical activity differently among individuals; it is unclear how these behaviours will evolve as the pandemic continues. In this observational study, dietary intake will be frequently collected using an artificial intelligence (AI)-enhanced mobile application combined with real-time analysis, and lifestyle behaviours from online questionnaires, to provide timely, relevant data for public health decision making.

DETAILED DESCRIPTION:
A thousand nine hundred and twenty adult men and women aged 18 years and older, living in the community and owning a smartphone or tablet, will be recruited all over Canada. Rapid recruitment will be achieved using social media and professional networks. All data will be collected online to allow a broad reach even in remote regions. Self-reported eating habits, physical activity, sleep, alcohol consumption, anxiety and depression data will be collected using validated questionnaires on an online survey platform, and dietary intake data using the mobile application Keenoa. With the application, participants take pictures of their meals, which are analyzed and accessible to researchers in real-time, providing comprehensive data on nutrient and food intake, and hence patterns and diet quality. Diet will be tracked for a full week at study entrance and repeated 6 times during a year, and once one year later, along with follow-up questionnaires on lifestyle behaviours.

The main study objectives are 1) to evaluate how eating habits, diet quality and related lifestyle behaviours of Canadian adults are impacted by confinement phases of the pandemic over one year; and 2) determine the association between eating behaviours and diet quality with contextual socio-demographic, education, emotional and health factors, and identify emerging explanatory factors as clusters.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years and over, living in Canada
* Owning a smartphone and having access to internet
* Able to read and understand English or French

Exclusion Criteria:

* Any active and uncontrolled acute disease that interferes with usual food intake
* Being hospitalized
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 1,920 adult men and women will be recruited from several regions of Canada, and stratified by age (18-45 y, 45-65 y, 65 y+).
Sampling Method: Non-Probability Sample
Enrollment: 2020 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Dietary intake | Two years
  Energy, macronutrients, micronutrients, and food intake assessed with the Keenoa mobile application

SECONDARY OUTCOMES:
Diet quality | Two years
  Calculated from food group intake as per the Canadian Healthy Eating Index
Eating habits | Two years
  Eating behaviors, food access and cooking skills collected from online questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University - School of Human Nutrition, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tessier AJ, Moyen A, Lawson C, Rappaport AI, Yousif H, Fleurent-Gregoire C, Lalonde-Bester S, Brazeau AS, Chevalier S. Lifestyle Behavior Changes and Associated Risk Factors During the COVID-19 Pandemic: Results from the Canadian COVIDiet Online Cohort Study. JMIR Public Health Surveill. 2023 Mar 30;9:e43786. doi: 10.2196/43786. PMID 36848226